CLINICAL TRIAL: NCT03526224
Title: Effect of Teriflunomide on Cortical Atrophy and Leptomeningeal Inflammation in Multiple Sclerosis: A Retrospective Observational Case-control Pilot Study
Brief Title: Teriflunomide Tecfidera LMCE
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director, Principal Investigator, University at Buffalo
Other Study IDs: STUDY00002359
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Tecfidera; Teriflunomide
MeSH Terms: interventions — Dimethyl Fumarate; teriflunomide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Aubagio: Individuals diagnosed with multiple sclerosis (MS) who have been treated with teriflunomide (Aubagio).
  Interventions: Drug: Teriflunomide
- Tecfidera: Individuals diagnosed with multiple sclerosis (MS) who have been treated with dimethyl fumarate (Tecfidera) and matched with the teriflunomide (Aubagio) patients on age, sex, disease duration, and disability level
  Interventions: Drug: Dimethyl Fumarate

INTERVENTIONS:
Drug: Dimethyl Fumarate — Individuals with MS treated with dimethyl fumarate (Tecfidera)
  Other Names: Tecfidera
  Groups: Tecfidera
Drug: Teriflunomide — Individuals with MS treated with teriflunomide (Aubagio)
  Other Names: Aubagio
  Groups: Aubagio

SUMMARY:
This study will investigate the effect of teriflunomide in reducing cortical gray matter (CGM) atrophy and leptomeningeal (LM) inflammation over 24 months compared to dimethyl fumarate (Tecfidera®)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS according to McDonald criteria
* Age 18-65 years
* Relapsing disease course
* Expanded Disability Status Scale (EDSS) score of ≤ 5.5
* MRI obtained at baseline (medication start date), 12 months, and 24 months
* Treated with 14mg of teriflunomide ≥ 3 months or with 240mg of dimethyl fumarate ≥ 3 months to meet inclusion, reflective of recommended dosing on the package label
* Clinical information available over the 24 month follow-up
* None of the exclusion criteria

Exclusion Criteria:

* Diagnosis of non-relapsing MS
* Use of experimental drug or investigational procedure during the study period
* Pregnancy during study period
* Severe hepatic impairment
* Relapse within 30 days prior to any of the 3 MRIs
* Corticosteroid use within 30 days prior to the MRIs
* Teriflunomide patients who have used leflunomide
* Pre-baseline use of alemtuzumab, cladribine, rituximab, or mitoxantrone
* Any other factor that, in the opinion of the investigator, would make the subject unsuitable for participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with MS who have used dimethyl fumarate or teriflunomide and had magnetic resonance imaging at baseline (before starting disease modifying therapy (DMT) in question), 12 months after starting DMT, and 24 months after starting DMT.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Percent change in CGM between teriflunomide and dimethyl fumarate | 24 months
  Percent change in cortical gray matter (CGM) between those on teriflunomide and dimethyl fumarate
LM CE lesions at 24 months | 24 months
  Frequency of leptomeningeal (LM) lesions as measured by presence (number) of LM contrast enhancing (CE) lesions foci on three-dimensional fluid-attenuated-inversion recovery (3D_FLAIR) MRI performed 10 minutes post-contrast injection between those on teriflunomide and dimethyl fumarate
CGM atrophy and LM inflammation | 24 months
  Association between the development of CGM atrophy and LM inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers

REFERENCES:
- [Result] Zivadinov R, Bergsland N, Carl E, Ramasamy DP, Hagemeier J, Dwyer MG, Lizarraga AA, Kolb C, Hojnacki D, Weinstock-Guttman B. Effect of Teriflunomide and Dimethyl Fumarate on Cortical Atrophy and Leptomeningeal Inflammation in Multiple Sclerosis: A Retrospective, Observational, Case-Control Pilot Study. J Clin Med. 2019 Mar 12;8(3):344. doi: 10.3390/jcm8030344. PMID 30870983